CLINICAL TRIAL: NCT05343507
Title: Complexity-enhancing Drugs to Treat Disorders of Consciousness (DoC): a Ketamine Study
Brief Title: Ketamine to Treat Patients With Post-comatose Disorders of Consciousness
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Centre Hospitalier Universitaire de Liege (Other); William Lennox Neurological Center UCLouvain (Unknown)
Responsible Party: Principal Investigator, Olivia Gosseries, Principal Investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021_211; 2021-002321-23 (EudraCT Number)
Record Dates: First submitted 2022-03-29; First posted 2022-04-25 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Disorder of Consciousness
Keywords: Psychedelics; Complexity; Ketamine; Clinical Diagnosis; Consciousness level
MeSH Terms: conditions — Consciousness Disorders | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, cross-over RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: One investigator not involved in the data acquisition and analysis, and the pharmacist who will prepare the syringe for the TCI will not be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketalar arm (Experimental): Patients will receive ketamine (sold in the form of Ketalar) intravenously, up to 0.75 µg/ml concentration, for a maximum of 90' minutes. Ketalar concentration will be increased slowly in a step-wise manner unless new signs of consciousness are evident.
  Interventions: Drug: Ketalar 50 MG/ML Injectable Solution
- Placebo arm (Placebo Comparator): Patients will receive placebo (saline solution)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketalar 50 MG/ML Injectable Solution — Intravenous solution (other info already provided)
  Other Names: Ketamine
  Arms: Ketalar arm
Drug: Placebo — Saline Solution
  Arms: Placebo arm

SUMMARY:
The investigators will run a Randomized Clinical Trial with 30 patients with disorders of consciousness (DoC), with intravenous subanesthetic doses of ketamine. Patients will simultaneously undergo TMS-EEG. The piloting will be done on 3 patients, with EEG only.

DETAILED DESCRIPTION:
The protocol will be organized in three phases: baseline, experimental, and follow-up. In the baseline, patients will receive a multimodal assessment [functional magnetic resonance imaging (fMRI), positron emission tomography (PET), electroencephalogram (EEG)]. The experimental phase is made of 2 sessions spaced 5 days apart: on day 1, patients will receive placebo (or ketamine), on day 5 patients will receive ketamine (or placebo). The order will be randomized and balanced. The investigators will use a targeted-controlled infusion (TCI) system to infuse a continuous subanesthetic dose of ketamine, which is known to have psychedelics effects, or a saline solution. The investigators will periodically assess for new signs of consciousness with the "simplified evaluation of consciousness disorders" (SECONDs) scale. The investigators will use transcranial magnetic stimulation coupled to EEG (TMS-EEG) to measure brain activity and calculate brain complexity. TMS-EEG will be performed from 20 minutes before the beginning of the infusion up to the max duration of the experiment (90 minutes). Another SECONDs will be performed on the following day of each session to control for carry-over effects. The primary outcomes are the emergence of new conscious behaviours and higher brain complexity following ketamine infusion. The secondary outcomes are baseline brain differences in neurophysiological and brain imaging measures between responders (new conscious behaviors or higher brain complexity) and non-responders (no new conscious behaviors or higher brain complexity). In the follow-up phase, patients' health will be evaluated at 1, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable
* Diagnosis of UWS or MCS based on repeated "coma recovery scale-revised) (CRS-R) or SECONDs
* More than 28 days post-insult
* Informed consent from the legal representative of the patient

Exclusion Criteria:

* Neurological medications other than anti-spasticity drugs in the last 2 weeks or 4 half-lives
* Previous neurological functional impairment other than related to their DoC
* A history of psychotic disorders
* Contraindication to MRI, EEG, PET or TMS
* Use of nitrates or other vasodilators, central nervous system acting agents such as barbiturates, morphine and related drugs.
* Use of drugs known to interact with ketamine (i.e., CYP3A4, diazepam, ...)
* Coronary insufficiency
* Other sympathomimetic drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
New conscious behaviours | Max 90 minutes from Ketamine Infusion
  New conscious behaviours (i.e., command following, visual pursuit) after the infusion of the ketamine as recorded via the "simplified evaluation of consciousness disorders" (SECONDs) behavioural scale, that are not seen before ketamine, during placebo infusion, or in baseline.
  The SECONDs has 8 items, with the most complex item linked to a higher conscious state. The score goes from 0 (coma) to 8 (emergent from the minimally conscious state).
Higher brain complexity | Max 90 minutes from Ketamine Infusion
  Higher brain complexity [perturbational complexity index (PCI) or Lempel-Ziv complexity (LZC)] during the infusion of ketamine. The investigators expect complexity to increase when new conscious behaviors are observed. If the patient does not show new signs of consciousness but has high complexity, the investigators expect to record memories of the experience in the follow-up phase.
  PCI and LZC values range from 0 (no complexity) to 1 (high complexity). The investigators expect complexity values to be proportional to the concentration of the drug.

SECONDARY OUTCOMES:
PET biomarker | From baseline
  Different baseline PET signal between responders (patients who show new signs of consciousness or higher brain complexity after the drug), and non-responders (who do not show new signs of consciousness or higher brain complexity). In particular, higher metabolism [measured by standardized uptake value (SUV)] in responders compared to non-responders.
MRI biomarker | From baseline
  Different baseline MRI between responders (patients who show new signs of consciousness or higher brain complexity after the drug), and non-responders (who do not show new signs of consciousness or higher brain complexity). In particular, higher resting-state BOLD activity in responders compared to non-responders and more preserved brain structures.
EEG power | From baseline
  Different baseline EEG signal between responders (patients who show new signs of consciousness or higher brain complexity after the drug), and non-responders (who do not show new signs of consciousness or higher brain complexity). In particular, higher alpha-band activity in responders compared to non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Gosseries, PhD, Principal Investigator — Coma Science Group (ULiege) & Centre du Cerveau2 (CHU Liege)
Locations (1):
- Centre Hospitalier Neurologique William Lennox, Ottignies-Louvain-la-Neuve, Wallonia, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymized and shared among collaborators upon reasonable request and agreement. If possible, data will be shared in an open-access database to ensure the values of open science.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be shared with collaborators for the specified time allocated to each respective project. Whereas, data shared on the database will be anonymized and available indefinitely.
Access Criteria: A written agreement between the groups (university or research teams)

REFERENCES:
- [Background] Casali AG, Gosseries O, Rosanova M, Boly M, Sarasso S, Casali KR, Casarotto S, Bruno MA, Laureys S, Tononi G, Massimini M. A theoretically based index of consciousness independent of sensory processing and behavior. Sci Transl Med. 2013 Aug 14;5(198):198ra105. doi: 10.1126/scitranslmed.3006294. PMID 23946194
- [Background] Scott G, Carhart-Harris RL. Psychedelics as a treatment for disorders of consciousness. Neurosci Conscious. 2019 Apr 21;2019(1):niz003. doi: 10.1093/nc/niz003. eCollection 2019. PMID 31024740